CLINICAL TRIAL: NCT04177082
Title: Evaluation of the Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-linking in Eyes With Corneal Thinning Conditions Using Peschke Riboflavin Solution
Brief Title: Safety and Effectiveness of the PXL-Platinum 330 System for CXL Using Riboflavin Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cornea Associates of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PXL-330-CAT
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Keratoconus; Pellucid Marginal Corneal Degeneration; Corneal Degeneration; Corneal Ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed 6mW/cm2 (Experimental): 6mW/cm2, with pulsed mode, 10 seconds on, 10 second off, for 30 minute total treatment time
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution
- Pulsed 4mW/cm2 (Experimental): 4mW/cm2, with pulsed mode, 10 seconds on, 10 second off, for 45 minute total treatment time
  Interventions: Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution

INTERVENTIONS:
Combination Product: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution — Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea
  Other Names: Corneal crosslinking

SUMMARY:
Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Collagen Cross-linking in Eyes With Corneal Thinning Conditions

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, pachymetry, and visual function.

ELIGIBILITY:
Inclusion Criteria

Subjects who have one or both eyes that meet criteria 1-4 and also meet at least 1 or more of criteria 5-11 will be considered candidates for this study:

1. 8 years of age or older
2. Signed written informed consent
3. Willingness and ability to comply with schedule for follow-up visits
4. Contact Lens Wearers Only:

   1. Removal of contact lenses for the required period of time prior to the screening refraction:

      Contact Lens Type Minimum Discontinuation Time Soft 3 days Soft Extended Wear 3 days Soft Toric 3 days Rigid gas permeable 2 Weeks
   2. Subjects who cannot function without wearing their contact lenses, may forgo discontinuation of contact lenses.
5. Presence of central or inferior steepening.
6. Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
7. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as:

   1. Fleischer ring
   2. Vogt's striae
   3. Decentered corneal apex
   4. Munson's sign
   5. Rizzutti's sign
   6. Apical Corneal scarring consistent with Bowman's breaks
   7. Scissoring of the retinoscopic reflex
   8. Crab-claw appearance on topography
8. Steepest keratometry (Kmax) value ≥ 47.20 D
9. I-S keratometry difference > 1.5 D on the Pentacam/Orbscan map or topography map
10. Posterior corneal elevation >16 microns
11. Thinnest corneal point >300 microns

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
K-Max | 12 Months
  Change in K-Max, compared to baseline
K-Mean | 12 Months
  Change in K-Mean, compared to baseline

SECONDARY OUTCOMES:
Uncorrected Visual Acuity | 12 Months
  Change in uncorrected visual acuity, compared to baseline
Best Corrected Visual Acuity | 12 Months
  Change in best corrected visual acuity, compared to baseline
Central Pachymetry | 12 Months
  Change in central pachymetry, compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tyrone McCall, MD, Principal Investigator — Cornea Associates of Texas
Locations (1):
- Cornea Associates of Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be held in a secure location. While summary outcomes data will be provided on request to other researchers and periodically at scientific conferences, protected health information will not.